CLINICAL TRIAL: NCT03209310
Title: The Effect of Trunk Control on Respiratory Muscle Strength and Activities of Daily Living in Children With Cerebral Palsy
Brief Title: The Effect of Trunk Control on Respiratory Muscle Strength
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Umut Apaydin, Gazi Ethical Committee, Gazi University
Other Study IDs: B.10.4.ISM.4.06.68.49/975
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Cerebral Palsy, Spastic; Posture; Respiratory Muscle Strength; Activities of Daily Living
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The children with Cerebral Palsy: Cerebral palsy (CP) can be defined as a group of disorders of movement and posture, causing activity limitation that are attributed to nonprogressive deficits that take place in the immature brain. The motor disorders of CP are often accompanied by deficits in sensation, cognition, communication, perception, behavioral and respiratory system.
- Control Group: Children with typical development were included in this study

SUMMARY:
Cerebral palsy (CP) can be defined as a group of disorders of movement and posture, causing activity limitation that are attributed to nonprogressive deficits that take place in the immature brain. The motor disorders of CP are often accompanied by deficits in sensation, cognition, communication, perception, behavioral and respiratory system .

Children with CP have many primary motor impairments such as selective mobility, muscle weakness, abnormal muscle tone, impaired coordination between agonist-antagonist muscles and insufficient postural control. These motor impairments also lead to secondary problems such as contractures and bone deformities. Whether primer or secondary, all these problems can reduce independence in activities of daily living (ADL) by affecting CP children at different levels.

There are several studies in children with CP that investigate the effects of trunk control and/or respiratory functions. However, there are very few studies examining the relationship of these functions which have direct effects on ADL. In these studies, the functions of children who are more heavily affected and unable to move have been examined. However, there are no studies examining the effect of trunk control on respiratory muscle strength in children with CP with a better mobility level. There are many factors affecting both trunk control and respiratory functions in these children. Therefore, in children with CP, who have better functional level and can move on their own, revealing the interaction between trunk control and respiratory functions may contribute significantly to the treatment process. For this reason, this study was planned to investigate the effect of trunk control on ADL and respiratory muscle strength in children with CP having a Gross Motor Functional Classification System (GMFCS) levels of 1 and 2 and to compare them with healthy children.

DETAILED DESCRIPTION:
Trunk control was evaluated by Trunk Control Measurement Scale (TCMS), ADL was evaluated by Pediatric Evaluation of Disability Inventory (PEDI) and respiratory muscle strength was evaluated by mouth pressure meter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP by a pediatric neurologist
* No significant scoliosis during postural evaluation
* Were having a level of 1 or 2 of GMFCS
* No orthopedic surgery or not having Botulinum Toxin-A injection in the last 6 months

Exclusion Criteria:

* Having speech or cooperative problems

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with Cerebral Palsy and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | 15 minutes
  TCMS measures the state of balance on the support surface and the ability to actively move body parts during functional activities, which are the two components of trunk control. TCMS consists of 15 items in total that are scored on 2, 3 or 4 point ordinal scale and administered bilaterally in case of clinical relevance. The total TCMS score ranges from 0 to 58. A high score on this scale represents a better performance

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | 30 minutes
  The ADLs of the children participating in the study were assessed by the Pediatric Evaluation of Disability Inventory (PEDI). It is a clinical measurement developed by Haley and used to evaluate the change in the functional skills, functional abilities and performance of children with disabilities. PEDI consists of two sections as Functional Skills Scale and Caregiver Assistance Scale. The first section, the Functional Skills Scale, is divided into three subscales: self-care, mobility and social function. This section, which consists of 197 items in total, is scored as unable (0) and capable (1). The second section of PEDI, the Caregiver Assistance Scale, is also divided into three subscales: self-care, mobility and social function. It consists of 20 items in total. Each item in this section is scored between 0 and 5. A score of 5 indicates that the child is completely independent, while a score of 0 indicates that the child is completely dependent on the caregiver.
Respiratory Muscle Strength | 15 minutes
  These measurements were made using the respiratory pressure meter (Micro Medical Micro RPM, UK) and performed according to American Thoracic Society/European Respiratory Society criteria (ATS. and ERS. 2002). Maximal Inspiratory Pressure (MIP) was measured in the residual volume after maximal expiration, while Maximal Expiratory Pressure (MEP) was measured in total lung capacity after maximum inspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Study Chair — Gazi U

IPD SHARING:
Plan to Share IPD: No